CLINICAL TRIAL: NCT05985551
Title: A Feasibility Study on the Timeframe of Superparamagnetic Iron Oxide Nanoparticles Administration in Patients Receiving Primary Systemic Therapy for Early Breast Cancer
Brief Title: Delayed SLND for Patients With Breast Cancer Undergoing Primary Systemic Treatment
Acronym: MagNeo
Status: Active, not recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Karakatsanis, Associate Professor, MD, PhD, Uppsala University
Other Study IDs: UUBreast03
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Chemotherapy Effect; Sentinel Lymph Node
Keywords: Neoadjuvant therapy; Breast Cancer; Superparamagnetic Iron oxide nanoparticles; SLND; Targeted axillary Dissection; Delayed SLND
MeSH Terms: conditions — Breast Neoplasms | interventions — ferric oxide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: SLND or TAD by the magnetic technique (SPIO) — All patients will receive Radioisotope according to standard of care. They will also receive SPIO in a timeframe of clinical convenience, depending on whether primary response is planned by means of MRI. For patients that are ycN0, SLND or TAD will be performed. For those that convert from cN1 to ycN0, the index lymph node will be marked with a paramagnetic marker. Axillary surgery will be undertaken with the magnetic technique and each retrieved lymph node will be controlled for radiation. Upon the completion of the procedure, a background control will be performed with the radioactive signal as guide, to ensure standard of care best practice. Any palpable lymph nodes that are not sentinels with either tracer may be removed at surgeon discretion but will be reported seperately.

SUMMARY:
The goal of this study was to assess the feasibility of SLND by superparamagnetic iron oxide nanoparticles (SPIO) in patients with early breast cancer planned for primary systemic therapy (PST) and whether this is affected by the timeframe of SPIO administration.

For this, patients with cN0/1 disease planned for PST received radioisotope as per routine on the day of surgery or the day before, and SPIO was injected in an extended timeframe, at any point from the day of surgery to before the induction of PST.

The main points to investigate are:

1. If the SPIO detection rate and concordance to the radiosotope are affected by time of SPIO injection
2. If the nodal yield and the accuracy of the procedure are affected

DETAILED DESCRIPTION:
Superparamagnetic Iron Nanoparticles (SPIO) have shown comparable performance to the standard of Radioisotope (RI) +/- blue dye (BD) for Sentinel Lymph Node Detection in breast cancer, with the advantage of clinical convenience due to easier accessibility, disposal and injection days before surgery.

More interestingly, SPIO provides the possibility for delayed SLND in the setting of a preoperative diagnosis of DCIS, enabling SLN detection weeks after breast surgery, only when specimen pathology has demonstrated invasive cancer, as shown in the SentiNot study. The role of SPIO for SLND in the setting of primary systemic therapy (PST) has not been extensively investigated, while the timeframe from SPIO administration to successful SLN detection in a similar fashion to SentiNot, but in the setting of PST has yet to been defined.

Current evidence suggest that RI-based SLN detection is the accepted standard following PST, with RI-based dual mapping specifically recommended in cN+-to-ycN0 patients, when SLND or targeted axillary dissection (TAD) are performed, as the number of SLNs retrieved has been inversely linked to the false negative rate of the procedure.

Apart from the logistic benefits of SPIO administration prior to PST, an aspect of potential interest is the ability to map the axilla, before the fibrotic changes induced by chemotherapy and lymphatic remodelling occur, that are a concern, especially in the node-positive patients at presentation.

However, in this case, it is imperative to investigate that SPIO remains detectable after a prolonged period of administration and that it does not migrate to higher nodal echelons. While preliminary data suggested feasibility, the aim of this dedicated study was to investigate the width of timeframe of SPIO administration in patients undergoing PST and how SPIO-based detection and concordance to the RI are affected.

In this study, patients scheduled for SLND or TAD after surgery will undergo the procedure with RI as the standard of care and will moreover receive SPIO. The administration of SPIO will take place either on the preoperative period but after the completion of PST, or before the induction of PST. The reason for this is to create a wide time-frame to allow for conclusion with regards to whether the mapping of the axilla prior PST by SPIO is a feasible technique that will then be addressed in a dedicated trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with non-metastatic primary breast cancer and cN0/cN1 axilla, as defined by clinical examination and axillary ultrasound (with fine needle aspiration or core biopsy verification of metastasis) intended for PST (chemotherapy, targeted treatment or endocrine therapy) with a curative intention at diagnosis,

Exclusion Criteria:

* Distant metastases at diagnosis
* Inflammatory breast cancer
* Tumor progression during PST for cN1 patients
* ycN1 after completion of PST
* surgery before the completion of PST for any reason (PST adverse effects, patient preference)
* cN1-to-ycN0 patients that opted for ALND

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that fulfilled all eligibility criteria as listed above
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between concordance (isotope and SPIO) and timepoint of SPIO administration to surgery | At surgery
  This endpoint is necessary in ensuring that prolonged SPIO administration does not result in the retrieval of "false" SLNs, in the case that SPIO migrates to higher nodal echelons. As the radioisotope is the current standard of care, the concordance of SPIO to the radioisotope and its correlation with time of SPIO adminstration is the appropriate surrogate endpoint.
Detection rate | At surgery
  The successful retrieval of at least one SLN detected by each tracer (SPIO or radioisotope) separately.
Concordance | At surgery
  The rate (patients with at least one SLN detected with both tracers/patients with at least one SLN detected with the radioisotope)

SECONDARY OUTCOMES:
Nodal yield | At surgery
  The median number of SLNs retrieved with each tracer
Nodal concordance | At surgery
  The rate (SLNs detected by both tracers/SLNs detected by the radioisotope)

OTHER OUTCOMES:
Detection rate for 2 and 3 SLNs | At surgery
  The successful retrieval of at least two and at least three SLN detected by each tracer (SPIO or radioisotope) separately.
Adverse events | From time of SPIO administration to four weeks after surgery
  Any adverse events reported in relation to SPIO administration

CONTACTS AND LOCATIONS:
Overall Officials: Andreas U Karakatsanis, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Patients have not been consented for IPD and separate consent should be sought for this. For any interest, contact andreas.karakatsanis@uu.se